CLINICAL TRIAL: NCT05425615
Title: Probing Language Processes Using Transcranial Magnetic Stimulation
Brief Title: Language Processing and TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Priyanka Shah-Basak, PhD, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 43228
Record Dates: First submitted 2022-06-07; First posted 2022-06-21 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Aphasia; Language
Keywords: TMS; Transcranial Magnetic Stimulation; Aphasia; Semantic processing; Phonological processing
MeSH Terms: conditions — Stroke; Aphasia; Language | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Multiple studies will be conducted in parallel. But within a study, the interventional assignment will be set to cross-over with 3-4 arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcomes assessor will both be blinded to intervention modalities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active TMS (Experimental): Deymed DuoMag XT-100 rTMS system (DM-XT100) connected to a 70-mm figure-of-eight coil with built-in cooling fans (also known as an air-cooled coil) will be used for delivering active repetitive or rapid TMS to the target site.
  Interventions: Device: Transcranial Magnetic Stimulation
- Control TMS (Active Comparator): Deymed DuoMag XT-100 rTMS system (DM-XT100) connected to a 70-mm figure-of-eight coil with built-in cooling fans will be used for delivering active repetitive or rapid TMS to the control site.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham TMS (Sham Comparator): Deymed DuoMag XT-100 rTMS system (DM-XT100) connected to a 70-mm figure-of-eight coil with built-in cooling fans will be used for delivering sham repetitive or rapid TMS to the control or target site.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Deymed DuoMag XT-100 rTMS
  Other Names: TMS

SUMMARY:
This study will examine the effect of TMS on people with stroke and aphasia as well as healthy individuals.

DETAILED DESCRIPTION:
To examine the brain's structure and specific language function and interactive relationships, investigators will implement repetitive or rapid TMS protocols in an active (or sham)-controlled, within-subject, randomized studies. Aims will evaluate the effects of short-term changes on each of the semantic or phonological language process of interest in isolation and changes in the interaction between language sub-processes and their interaction with other cognitive domains that directly or indirectly affect language functions. The brain targets for TMS application will be informed by existing evidence on (correlational but not causal) associations between language regions and specific language processes from numerous prior neuroimaging (e.g., functional magnetic resonance imaging or fMRI) and neuropsychological studies. Healthy individuals and/or stroke survivors with aphasia will be recruited to address these aims.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with left hemisphere stroke
* Consent date >= 1 month after stroke onset
* Right-handed
* Fluent in English
* 18 years of age or older

Exclusion Criteria:

* Severe cognitive, auditory or visual impairments that would preclude cognitive and language testing
* Non-decisional per decisionality questionnaire or other clinical assessment
* Presence of major untreated or unstable psychiatric disease (e.g. schizophrenia, bipolar disease)
* A chronic medical condition that is not treated or is unstable
* Presence of

  1. cardiac stimulators or pacemakers or intracardiac lines
  2. neurostimulators
  3. medication infusion device
  4. any other implants near the scalp (e.g., cochlear implants) or in the eye
  5. metal in the body
* Pregnancy
* History of skull fractures, or skin diseases
* History of ongoing or unmanaged seizures or a family history of epilepsy
* Presence of factors that potentially decrease seizure thresholds
* On pro-convulsant medications
* Untreated Sleep deprivation or insomnia
* Ongoing alcoholism or illegal drug abuse (e.g., cocaine or MDMA users)
* History of dyslexia or other developmental learning disabilities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Reaction time on language task performance | Language tasks administered immediately before and/or after TMS administration (same day).
  Improvement on language task performance as measured by decrease in reaction time.
Accuracy on language task performance | Language tasks administered immediately before and/or after TMS administration (same day).
  Improvement on language task performance as measured by increase in accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Shah-Basak, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Devlin JT, Watkins KE. Stimulating language: insights from TMS. Brain. 2007 Mar;130(Pt 3):610-22. doi: 10.1093/brain/awl331. Epub 2006 Nov 29. PMID 17138570
- [Background] Epstein CM. Transcranial magnetic stimulation: language function. J Clin Neurophysiol. 1998 Jul;15(4):325-32. doi: 10.1097/00004691-199807000-00004. PMID 9736466
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. Brain Lang. 2011 Jul;118(1-2):40-50. doi: 10.1016/j.bandl.2011.02.005. Epub 2011 Apr 2. PMID 21459427
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Keel JC, Smith MJ, Wassermann EM. A safety screening questionnaire for transcranial magnetic stimulation. Clin Neurophysiol. 2001 Apr;112(4):720. doi: 10.1016/s1388-2457(00)00518-6. No abstract available. PMID 11332408
- [Background] Lehtinen H, Makela JP, Makela T, Lioumis P, Metsahonkala L, Hokkanen L, Wilenius J, Gaily E. Language mapping with navigated transcranial magnetic stimulation in pediatric and adult patients undergoing epilepsy surgery: Comparison with extraoperative direct cortical stimulation. Epilepsia Open. 2018 Apr 6;3(2):224-235. doi: 10.1002/epi4.12110. eCollection 2018 Jun. PMID 29881801
- [Background] Lerner AJ, Wassermann EM, Tamir DI. Seizures from transcranial magnetic stimulation 2012-2016: Results of a survey of active laboratories and clinics. Clin Neurophysiol. 2019 Aug;130(8):1409-1416. doi: 10.1016/j.clinph.2019.03.016. Epub 2019 Apr 6. PMID 31104898
- [Background] Narayana S, Gibbs SK, Fulton SP, McGregor AL, Mudigoudar B, Weatherspoon SE, Boop FA, Wheless JW. Clinical Utility of Transcranial Magnetic Stimulation (TMS) in the Presurgical Evaluation of Motor, Speech, and Language Functions in Young Children With Refractory Epilepsy or Brain Tumor: Preliminary Evidence. Front Neurol. 2021 May 19;12:650830. doi: 10.3389/fneur.2021.650830. eCollection 2021. PMID 34093397
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Pascual-Leone A, Bartres-Faz D, Keenan JP. Transcranial magnetic stimulation: studying the brain-behaviour relationship by induction of 'virtual lesions'. Philos Trans R Soc Lond B Biol Sci. 1999 Jul 29;354(1387):1229-38. doi: 10.1098/rstb.1999.0476. PMID 10466148
- [Background] Pascual-Leone A, Walsh V, Rothwell J. Transcranial magnetic stimulation in cognitive neuroscience--virtual lesion, chronometry, and functional connectivity. Curr Opin Neurobiol. 2000 Apr;10(2):232-7. doi: 10.1016/s0959-4388(00)00081-7. PMID 10753803
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A. Screening questionnaire before TMS: an update. Clin Neurophysiol. 2011 Aug;122(8):1686. doi: 10.1016/j.clinph.2010.12.037. Epub 2011 Jan 11. No abstract available. PMID 21227747
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Rossini PM, Rossi S. Clinical applications of motor evoked potentials. Electroencephalogr Clin Neurophysiol. 1998 Mar;106(3):180-94. doi: 10.1016/s0013-4694(97)00097-7. PMID 9743275
- [Background] Shrout PE, Rodgers JL. Psychology, Science, and Knowledge Construction: Broadening Perspectives from the Replication Crisis. Annu Rev Psychol. 2018 Jan 4;69:487-510. doi: 10.1146/annurev-psych-122216-011845. PMID 29300688
- [Background] Walsh V, Cowey A. Transcranial magnetic stimulation and cognitive neuroscience. Nat Rev Neurosci. 2000 Oct;1(1):73-9. doi: 10.1038/35036239. PMID 11252771
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Wilson SM, Eriksson DK, Schneck SM, Lucanie JM. A quick aphasia battery for efficient, reliable, and multidimensional assessment of language function. PLoS One. 2018 Feb 9;13(2):e0192773. doi: 10.1371/journal.pone.0192773. eCollection 2018. PMID 29425241